CLINICAL TRIAL: NCT03312283
Title: A Randomized, Double-blind, Two-group Parallel, Positive-controlled Clinical Phase I Trial Comparing the Safety, Pharmacokinetics and Pharmacodynamics of QL1205 and Lucentis® in Patients With Wet Age-related Macular Degeneration.
Brief Title: Evaluating of the Safety, Pharmacokinetics and Pharmacodynamics of QL1205 and Lucentis® in Patients With Wet AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QL1205-001
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2017-10

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1205 (Experimental): QL1205 injection (0.5mg) by vitreous injection once a month for three months（D1、D29、D57）
  Interventions: Drug: QL1205
- Lucentis (Active Comparator): Lucentis® injection(0.5mg) by vitreous injection once a month for three months（D1、D29、D57）
  Interventions: Drug: lucentis

INTERVENTIONS:
Drug: lucentis — intravitreal injection of 0.5 mg (0.05 ml), Q4W, continuous administration for 3 times (D1, D29, D57)
  Other Names: Ranibizumab Injection
  Arms: Lucentis
Drug: QL1205 — intravitreal injection of 0.5 mg (0.05 ml), Q4W, continuous administration for 3 times (D1, D29, D57)
  Other Names: Ranibizumab Injection
  Arms: QL1205

SUMMARY:
This is a randomized, double-blind, two-group parallel, positive-controlled clinical Phase I trial comparing the safety, pharmacokinetics and pharmacodynamics of QL1205 and Lucentis® in patients with wet age-related macular degeneration.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind, two-group parallel, positive-controlled clinical trial at four centers.

The primary objective is to assess the initial clinical safety of intravitreal injection of QL1205 or Lucentis® in patients with wet age-related macular degeneration (wet-AMD).

The secondary objective are to assess the initial clinical effectiveness and pharmacokinetic characteristics of intravitreal injection of QL1205 or Lucentis® in patients with wet age-related macular degeneration (wet-AMD).

Subjects would sequentially enrolled according to the protocol in one of two cohorts.Subjects would receive a single 0.5mg of QL1205 or Lucentis® once a month for three months through vitreous injection.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form, and willing to receive follow-up according to the time stipulated by the trial;
2. Aged ≥50 years or ≤80 years, male or female (including the boundary value);
3. The target eye must meet the following requirements; Has newly occurring or relapsed subfoveal and perifoveal active choroidal neovascularization (CNV) lesions secondary to AMD; The total area of all types of lesions is ≤30 mm2(the area of 12 optic discs); The best corrected visual acuity is 78-19 letters (equivalent to Snellen visual acuity of 20/32 to 20/400); No refractive media opacity or myosis affecting fundus examination;
4. The best corrected visual acuity of the subject's non-target eye is ≥19 letters (equivalent to Snellen visual acuity of 20/400).

Note: If the subject's eyes both meet the inclusion criteria, the investigator will determines the target eye from a medical point of view.

Exclusion Criteria:

Patients with any of the following eye conditions:

1. The investigator judges that the target eye is currently suffering or used to suffer from non-exudative AMD disease affecting macular detection, or ocular diseases affecting central visual acuity (including central venous obstruction, diabetic retinopathy, uveitis, vascular striation, pathological myopia, retinal detachment, macular hole, etc.);
2. The target eye's CNV is secondary to diseases other than AMD, such as trauma, pathological myopia,etc.;
3. Either eye has previously received drug treatment for CNV (e.g., Lucentis, Avastin, Eylea, Composin, Acaconac, triamcinolone, steroids, etc.)
4. The target eye has subretinal hemorrhage, and hemorrhagic area is ≥ 50% of the total area of the lesion, or the subfoveal bleeding area is ≥ 1 optic disc area;

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of QL1205 | 85 days
  To evaluate the safety of QL1205, compared to that of Lucentis (registered trademark) in patients with neovascular AMD.This will be done by assessment of vital signs, physical examination, laboratory blood tests and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Xu, professor, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; mingwei zhao, professor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No